CLINICAL TRIAL: NCT01390259
Title: Hypoglycemia Prevention After Exercise in Adolescent T1DM Patients Using a Control to Range System
Acronym: MDB005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Abbott Diabetes Care (Industry); DexCom, Inc. (Industry); Insulet Corporation (Industry); University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Marc Breton, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14758
Record Dates: First submitted 2011-07-06; First posted 2011-07-11 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed Loop Control (CLC) (Experimental): The CLC used a computer to make recommendations for their insulin treatment. This study arm was designed to demonstrate management of glucose using a modular insulin management system based on continuous glucose monitoring and targeted towards the avoidance of hypoglycemic and prolonged hyperglycemic episodes (i.e. control to range). This system was designed to both:
  * monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  * predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Interventions: Device: Closed-Loop
- Open Loop (Placebo Comparator): The subject were in charge of their insulin treatment.
  Interventions: Device: Open-Loop

INTERVENTIONS:
Device: Open-Loop — This admission was to assess the subjects' level of glucose control and created a base to compare the performance of the closed-loop system. Subjects monitored their own blood glucose values and administer their basal/bolus as they would at home. Otherwise, the admission remained the same as in the closed-loop admission (i.e. meals, exercise, etc...).
  Arms: Open Loop
Device: Closed-Loop — In this study, the researchers compared the management of diabetes during physical activity and meals with the closed-loop system developed at the University of Virginia. This system uses two DexComTM Seven Continuous Glucose Monitor, a computer containing an investigational control algorithm (well-defined instructions that are expressed in mathematical equations), and an OmniPod Insulin Management System, a portable subcutaneous (under the skin) insulin pump. During the closed-loop admission, the computer based algorithm used CGM values to make recommendations of insulin treatment. The study included a challenge to the insulin management system with meals and mild exercise, so as to demonstrate its capacity to avoid large glucose excursion with changing metabolic state.
  Arms: Closed Loop Control (CLC)

SUMMARY:
In this protocol the investigators plan to demonstrate management of glucose using a modular insulin management system based on continuous glucose monitoring and targeted towards the avoidance of hypoglycemic and prolonged hyperglycemic episodes (i.e. control to range). The protocol is designed to challenge the insulin management system with meals and mild exercise, so as to demonstrate its capacity to avoid large glucose excursion with changing metabolic state. This system is designed to both

* monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
* predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.

The investigators plan to enroll 12 adolescent T1DM patients (expected retention 10/12) and compare glucose control performances under two treatments: standard vs. the new insulin management system. The protocol will include a total of 5 admissions per subject (3 out-patients and 2 in-patients): screening, CGM insertion 1, CGM insertion 2, inpatient 1 and inpatient 2. During the 24h inpatient admissions the patients will be challenged with 30 minutes of mild exercise and 3 meals, insulin coverage of these events will vary depending on the chosen treatment, each subject will be exposed to both studied treatments (repeated measure design). The order of treatment during the inpatient admissions will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age and up to and including 18 years of age.
* Have type 1 diabetes mellitus as defined by American Diabetes Association criteria or judgment of physician for at least 1 year (including those who may also be treated with metformin).
* Use of an insulin pump
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study
* Willingness to use lispro (Humalog) insulin for the duration of the inpatient study
* Demonstration of proper mental status and cognition for the study
* Willingness to stop using any dietary supplements for two weeks prior to admission and for the duration of their participation
* HemoglobinA1c < 10.0
* A score of 2 or greater on the hypoglycemia unawareness scale, see Attachment A
* Tanner Stage II or greater (not pre-pubertal) on screening physical exam
* Body weight of 30 kg or more at screening
* BMI must be under 95th percentile for age based on published BMI reference standards

Exclusion Criteria:

* Age <12 or >18
* Pregnancy
* Hematocrit <37% (females); <36% (males)
* HemoglobinA1c ≥ 10.0
* Any symptomatic coronary artery disease, or a history of congenital heart abnormalities.
* Score of less than 2 on the hypoglycemia unawareness scale
* Tanner Stage I on screening physical exam
* Use of a medication that significantly lowers heart rate (beta blockers, reserpine, guanethidine, methyldopa, clonidine, cimetidine, digitalis, calcium channel blockers, amiodarone, antiarrythmic drugs, or lithium)
* Congestive heart failure
* History of a cerebrovascular event
* Use of a medication that significantly impacts glucose metabolism (oral steroids)
* Atrial fibrillation
* Uncontrolled hypertension (resting blood pressure >140/90)
* History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the FreeStyle NavigatorTM CGM or DexCom Seven® (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
* Active enrollment in another clinical trial
* Allergy or adverse reaction to lispro insulin
* Known adrenal gland problem, pancreatic tumor, or insulinoma
* Current alcohol abuse by patient history, substance abuse by patient history, or severe mental illness
* Retinopathy and renal failure
* Uncontrolled anxiety or panic disorder
* Known bleeding diathesis or dyscrasia
* Renal insufficiency (creatinine >1.5)
* Any comorbid condition affecting glucose metabolism
* Body weight of less than 30 kg at screening
* BMI equal to or greater than 95th percentile for age based on published BMI reference standards. See Appendix B.
* Asthma or exercise -induced asthma
* Any mobility-restrictive condition
* Children who are wards of state or at high risk for becoming wards of state

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc D. Breton, Ph.D., Principal Investigator — University of Virginia, Center for Diabetes Technology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Breton M, Farret A, Bruttomesso D, Anderson S, Magni L, Patek S, Dalla Man C, Place J, Demartini S, Del Favero S, Toffanin C, Hughes-Karvetski C, Dassau E, Zisser H, Doyle FJ 3rd, De Nicolao G, Avogaro A, Cobelli C, Renard E, Kovatchev B; International Artificial Pancreas Study Group. Fully integrated artificial pancreas in type 1 diabetes: modular closed-loop glucose control maintains near normoglycemia. Diabetes. 2012 Sep;61(9):2230-7. doi: 10.2337/db11-1445. Epub 2012 Jun 11. PMID 22688340

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Loop First, Then Closed-Loop: Open-Loop first, then Closed-Loop control (CLC)
  Experimental, CLC admission: The CLC used a computer to make recommendations for their insulin treatment. This system was designed to both:
  1. monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  2. predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Placebo Comparator: Open Loop admission. The subjects were in charge of their insulin treatment.
- Closed-Loop Control First, Then Open-Loop: Closed-Loop control (CLC) first, then Open-Loop
  Experimental, CLC admission: The CLC used a computer to make recommendations for their insulin treatment. This system was designed to both:
  1. monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  2. predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Placebo Comparator: Open Loop admission. The subjects were in charge of their insulin treatment.
Period: Overall Study
Arm/Group | Open-Loop First, Then Closed-Loop | Closed-Loop Control First, Then Open-Loop
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Adolescents: Adolescents participated in both the Standard Control to Range (sCTR) Closed-Loop Control (CLC) Admission and the Open-Loop admission.
  Experimental: The CLC used a computer to make recommendations for their insulin treatment. This system was designed to both:
  1. monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  2. predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Placebo Comparator: Open Loop. The subjects were in charge of their insulin treatment.
Arm/Group | Adolescents
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
HbA1c [Mean (Standard Deviation); unit: percent] — Glycated hemoglobin
  percent | 8.6 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemic Events
Description: Number of hypoglycemic events below 70 mg/dL per patient per day
  Hypoglycemic event is defined as consecutive YSI plasma glucose measurements below 70 or moderate hypoglycemic symptoms
Time Frame: 22 hours
Measure: Mean (Standard Error); unit: events/patient
Groups:
- Closed-Loop Control (CLC): The CLC used a computer to make recommendations for their insulin treatment. This study arm was designed to demonstrate management of glucose using a modular insulin management system based on continuous glucose monitoring and targeted towards the avoidance of hypoglycemic and prolonged hyperglycemic episodes (i.e. control to range). This system was designed to both:
  * monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  * predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Closed-Loop: During the closed-loop admission, the computer based algorithm used CGM values to make recommendations of insulin treatment. Standard Control to Range (sCTR).
- Open-Loop: The subjects were in charge of their insulin treatment.
  Open-Loop: This admission was to assess the subjects' level of glucose control and created a base to compare the performance of the closed-loop system. Subjects monitored their own blood glucose values and administer their basal/bolus as they would at home. Otherwise, the admission remained the same as in the closed-loop admission (i.e. meals, exercise, etc...).
Arm/Group | Closed-Loop Control (CLC) | Open-Loop
Number analyzed (Participants) | 11 | 11
events/patient
  Overall (t=22h) | 0.27 (0.19) | 1.0 (0.5)
  Exercise (t=0.5h) | 0.18 (0.12) | 0.18 (0.12)
  Recovery (t=1h) | 0 (0) | 0.18 (0.12)
  Overnight (t=7h) | 0 (0) | 0.18 (0.18)

2. Secondary Outcome: Percent Time in Euglycemia
Description: Percent of time the patient plasma glucose as measured by YSI is between 70mg/dl and 180mg/dl
Time Frame: 22 hours
Measure: Mean (Standard Error); unit: percentage of time in range
Arm/Group | Closed-Loop Control (CLC) | Open-Loop
Number analyzed (Participants) | 11 | 11
percentage of time in range
  Overall (t=22h) | 65.1 (6.8) | 50.2 (9.7)
  Day (t=15h) | 74.0 (5.2) | 57.0 (8.9)
  Night (t=7h) | 56.0 (11.8) | 43.6 (13.3)

3. Secondary Outcome: Mean Glucose
Description: Average plasma glucose concentration in mg/dl
Time Frame: 22 hours
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Closed-Loop Control (CLC) | Open-Loop
Number analyzed (Participants) | 11 | 11
mg/dL
  Overall (t=22h) | 166.24 (7.23) | 176.1 (18.04)
  Day (t=15h) | 155.44 (7.76) | 160.57 (16.54)
  Night (t=7) | 177.29 (8.23) | 193.04 (22.08)

ADVERSE EVENTS:
Arm/Group | Adolescents
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes